CLINICAL TRIAL: NCT01959659
Title: A Non-Interventional Study of Patients With Persistent Symptoms of Schizophrenia to Describe Medical Resource Utilization and Burden of Illness
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MN28222
Record Dates: First submitted 2013-09-26; First posted 2013-10-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This non-interventional, cross-sectional survey and retrospective review will evaluate the medical resource utilization and burden of illness in patients who have persistent symptoms of schizophrenia despite receiving adequately dosed antipsychotic treatment and who have not had an acute exacerbation in the 3 months prior to enrolment. Medical records will be reviewed for a minimum of 3 months and up to 12 months prior to screening. Data collection at a single visit will include rating scales and questionnaires that reflect the clinical status and the quality of life of the patients and the economic impact of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients who have a clinical diagnosis of schizophrenia as documented in their medical records
* Patients who, in the opinion of the investigator, have had on-going, persistent symptoms of schizophrenia for at least the last 3 months prior to enrolment
* Patients who, in the opinion of the investigator, have been prescribed adequate doses of antipsychotic treatment for at least the last 3 months
* Patient has adequate spoken local language

Exclusion Criteria:

* Acute exacerbation of schizophrenia within the last 3 months prior to enrolment
* Enrolment in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent symptoms of schizophrenia despite receiving adequately dosed antipsychotic treatment and who have not had an acute exacerbation in the last 3 months
Sampling Method: Probability Sample
Enrollment: 1431 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Medical resource utilization (in-/out-patient hospital services, community-based day service, other health care contacts) of patients with persistent symptoms of schizophrenia | in the 3 to 12 months prior to screening

SECONDARY OUTCOMES:
Level/severity of schizophrenia symptoms: Clinical rating scales scores (PANSS, CGI-S, PSP, WoRQ, NSA-4, HoNOS) | Observational visit Day 1
Patient health-related quality of life (HRQoL) questionnaires | Observational visit Day 1
Caregiver's burden as assessed by questionnaires | Observational visit Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (95):
- Australia (2):
  - Epping, New South Wales
  - Everton Park, Queensland
- Czechia (8):
  - Brno
  - Brno, Jihormoravsky Kraj
  - Hradec Králové
  - Olomouc
  - Pilsen
  - Prague
  - Praha 8 - Bohnice
  - Přerov
- France (23):
  - Bohars
  - Bron
  - Brumath
  - Colombes
  - Digne-les-Bains
  - Fitz-James
  - Hénin-Beaumont
  - Leyme
  - Lille
  - Montauban
  - Montpellier
  - Neuilly-sur-Marne
  - Novillars
  - Paris
  - Poitiers
  - Pontarlier
  - Provins
  - Reims
  - Rennes
  - Saint-Égrève
  - Saint-Nazaire
  - Sens
  - Verdun
- Italy (23):
  - Chieti, Abruzzo
  - L’Aquila, Abruzzo
  - Aosta, Aosta Valley
  - Foggia, Apulia
  - Roggiano Gravina, Calabria
  - Salerno, Campania
  - Solofra, Campania
  - Bologna, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Legnago, Lombardy
  - Monza, Lombardy
  - Pieve di Coriano, Lombardy
  - Varese, Lombardy
  - Campobasso, Molise
  - Novara, Piedmont
  - Adrano, Sicily
  - Lido di Camaiore, Tuscany
  - Pisa, Tuscany
  - Siena, Tuscany
- Russia (9):
  - Kemerovo
  - Lipetsk
  - Moscow
  - Moscow Region
  - Nizhny Novgorod
  - Petrozavodsk
  - Saint Petersburg
  - Samara
  - Talagi
- Spain (22):
  - Almería, Almeria
  - Manacor, Balearic Islands
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Santander, Cantabria
  - Torrelavega, Cantabria
  - A Coruña, La Coruña
  - Alcalá de Henares, Madrid
  - Arganda, Madrid
  - Madrid, Madrid
  - Majadahonda, Madrid
  - Málaga, Malaga
  - Pamploma, Navarre
  - Mos, Pontevedra
  - Vigo, Pontevedra
  - Langreo, Principality of Asturias
  - Dos Hermanas, Sevilla
  - Reus, Tarragona
  - Toledo, Toledo
  - Valencia, Valencia
  - Vitoria-Gasteiz, Vizcaya
  - Zaragoza, Zaragoza
- Turkey (Türkiye) (8):
  - Ankara
  - Diyarbakır
  - Gaziantep
  - Istanbul
  - Kocaeli
  - Manisa
  - Mersin
  - Samsun